CLINICAL TRIAL: NCT00497627
Title: Quality of Life and Cardiometabolic Risk Factors in Patients After Debanding
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Cantonal Hospital, Frauenfeld (Other)
Responsible Party: Principal Investigator, Markus Mueller, PD Dr. med., University of Zurich
Other Study IDs: StV 38-2006
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Bariatric Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Follow up of debanding patients

DETAILED DESCRIPTION:
Follow up of debanding patients regarding cardiometabolic risk factors

ELIGIBILITY:
Inclusion criteria:

* Previous debanding after lap. gastric bypass

Exclusion criteria:

* Further bariatric procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Follow up of debanding patients regarding cardiometabolic risk factors
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2007-01; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 2 to 5 years after debanding

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland